CLINICAL TRIAL: NCT03808766
Title: A Study on the Angioarchitecture of Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VIR-18-09
Record Dates: First submitted 2018-10-10; First posted 2019-01-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: Tumors are categorized into 3 groups based on the longest diameter of the largest tumor:
  Group 1: ≤3cm Group 2: >3cm to 7cm Group 3: >7cm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tumor <=3cm (Other): Embolization with particulate or liquid embolic agent
  Interventions: Other: embolization
- Tumor >3cm to 7cm (Other): Embolization with particulate or liquid embolic agent
  Interventions: Other: embolization
- Tumor > 7cm (Other): Embolization with particulate or liquid embolic agent
  Interventions: Other: embolization

INTERVENTIONS:
Other: embolization — Patient with a diagnosis of HCC and a treatment plan to receive partial hepatectomy will receive transarterial embolization under local anesthesia 2 weeks before the surgery. Angiographic examinations of the tumor before and after embolization of the tumor will be performed. Histological examination of the tumor in the surgical specimens will be performed.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the commonest solid malignancies in Hong Kong as well as globally. Transarterial therapy has been playing an important role in the treatment algorithm for patients with HCC. The primary purpose of transarterial therapy is eradication of the viability of the targeted tumors. The treatment outcomes have been variable among the various treatments, in general, there is still much room for improvement, especially for large size tumors. From the studies on Transarterial chemoembolization (TACE), it is known that the treatment outcome is affected by the nature and the formulation of therapeutic agents that are delivered, which is related to the angioarchitecture of the tumor. Knowledge on the angioarchitecture of HCC is essential for the understanding of the requirements for effective transarterial treatment of HCC. This prospective study is aimed to study the angioarchitecture of HCC.

DETAILED DESCRIPTION:
Embolization is performed within 2 weeks before the scheduled date of partial hepatectomy. The purpose of the timing is two folded, it allows observation of the embolization effect to be differentiated among the various embolic agents, it also allows time for the patient and the liver to recover from the embolization.

The patient then receives partial hepatectomy within 2 weeks unless the result of liver function tests shows contraindication to surgery, in which case the liver function test is further evaluated on a weekly basis until the findings are acceptable, and surgery is scheduled accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. HCC suitable for partial hepatectomy
3. Child-Pugh A or B cirrhosis
4. Eastern Cooperative Oncology Group performance score 0 or 1
5. Barcelona clinic liver cancer (BCLC) staging A or B
6. HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology
7. Massive expansive tumor morphology with measurable lesion on CT (characterized by well-defined spherical or globular configuration, with or without tumor capsule or satellite lesions)

Exclusion Criteria:

1. Previous treatment with liver resection, ablation, chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy),
2. Evidence of tumor invasion of portal vein or hepatic vein
3. History of acute tumor rupture presenting with hemo-peritoneum
4. Infiltrative tumor morphology (characterized by ill- defined tumor margin and amorphous configuration) or diffuse tumor morphology (characterized by large number of small nodules)
5. Serum creatinine level > 150umol/L

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
arterial flow through the tumor | within one hour
  Digital subtraction angiography (DSA) is performed before and after embolization, through catheterization of the arterial branches supplying the tumor, images from arterial phase to delayed phase are captured. Contrast distribution at the arterial tumor branches, arterioles, tumor sinusoids, peri-tumoral liver, and peri-tumoral portal venules are observed.

SECONDARY OUTCOMES:
The degree of tumor necrosis | within 2 weeks after embolization
  The percentage of viable residual HCC is assessed quantitatively in increments of 5 %, with the measurement of the largest axial diameter of viable HCC compared to that of the whole tumor using a microscopic ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No